CLINICAL TRIAL: NCT00495339
Title: Multicenter Open Non-Comparative Clinical Study to Evaluate the Efficacy and Safety of Three Months TAVANIC Course (Levofloxacin) in Combine Treatment of Multi-Drug-Resistant Tuberculosis (MDR-TB)
Brief Title: MDR TB, Levofloxacin, Multi-Drug-Resistant Pulmonary Tuberculosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEVOF_L_00972
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2008-06

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Levofloxacin

ARMS (1):
- 1 (Experimental): Levofloxacin
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin — 500-1000 mg once a day daily per os with combination of drugs.

SUMMARY:
Estimate of clinical and microbiological efficacy of Levofloxacin (Tavanic) in combine therapy of MDR TB.

Estimate of safety of Levofloxacin (Tavanic) in combine therapy of MDR TB.

ELIGIBILITY:
Inclusion Criteria:

* Drug-resistant pulmonary tuberculosis laboratory diagnosed

Exclusion Criteria:

* Known hypersensitivity to levofloxacin, other quinolones
* Patient with epilepsy and central nervous system diseases
* Renal insufficiency with serum creatinine lower than 50 ml/min
* Arterial hypertension, ischemic heart disease in acute phase
* Gastro-intestinal diseases, liver diseases in acute phase
* History of drug and alcohol abuse
* Patient with history of tendon disorders related to fluoroquinolone administration
* Pregnancy and breast-feeding women
* Immune system disorders related to chemotherapy, AIDS, long term administration of corticosteroids

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with bacterioexcretion | 1 month, 2 months, 3 months
Dynamics of chest radiograph | 3 months
Dynamics of Intoxication | 1 month, 2 months, 3 months
All clinical and laboratory adverse events | from the signature of the Informed Concent Form (ICF) up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Marina Atarshchikova, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Moscow, Russia